CLINICAL TRIAL: NCT03713177
Title: Awareness and Knowledge of Systemic Diseases and Its Relevance to Oral Health Care Among Dentists and Dental Interns: Observational Cross-sectional Study
Brief Title: Awareness of Systemic Diseases and Its Dental Implications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelaziz Mohamed Ahmed Moussa, Postgraduate Student, Cairo University
Other Study IDs: Med159
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Dental Awareness of the Relation Between Systemic Disease and Oral Health Conditions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ministry of health - Cairo: Dentists working for Egyptian ministry of health - Cairo
- Interns: Dental interns of Cairo University

SUMMARY:
Implications of systemic diseases on Oral health and their manifestation

DETAILED DESCRIPTION:
Systemic Diseases have oral manifestations and these oral manifestation may affects the treatment plan and may affect the drugs given after dental treatment hence the study aims to assess the awareness and knowledge of systemic diseases and its implications in the dental field

ELIGIBILITY:
Inclusion Criteria:

* Dentists working for Egyptian ministry of health - Cairo.
* Dental interns of Cairo University.

Exclusion Criteria:

* Those who refused to share information.
* Candidates who refused to sign consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dental health care providers in different settings
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
degree of awareness among dentists and dental students about systemic diseases and its relevance to oral health. | 1 Year
  Questionnaire

SECONDARY OUTCOMES:
Assess their knowledge about dental management of these cases | 1 year
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Abdelaziz Moussa, Graduate, Principal Investigator — Post grad Student at Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tavares M, Lindefjeld Calabi KA, San Martin L. Systemic diseases and oral health. Dent Clin North Am. 2014 Oct;58(4):797-814. doi: 10.1016/j.cden.2014.07.005. Epub 2014 Aug 7. PMID 25201543